CLINICAL TRIAL: NCT05301686
Title: Is There a Correlation Between Surgical Technique for Primary Anterior Cruciate Ligament Surgery and the Risk of Subsequent Formation of Fibrous Cyst (Cyclops) in the Knee Joint, Which Leads to the Need for Surgical Removal of the Cyclops? A Registry Study With Patients Operated on With Cruciate Ligament Reconstruction at Aarhus University Hospital From 2005-2019.
Brief Title: Is There a Correlation Between Surgical Technique for Primary Anterior Cruciate Ligament Surgery and the Risk of Subsequent Formation of Fibrous Cyst (Cyclops) in the Knee Joint, Which Leads to the Need for Surgical Removal of the Cyclops?
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Other Study IDs: EC: 1-10-72-274-21
Record Dates: First submitted 2022-03-20; First posted 2022-03-31 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cyclop Arthrofibrosis Anterior Cruciate Ligament

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Cyclop lesion: Patients with an anterior cruciate ligament reconstruction with a symptomatic Cyclop lesion leading to a arthroscopy within 2 years after primary surgery
  Interventions: Procedure: Patients with Cyclop lesion
- Patients without Cyclop lesion: Patients without no arthroscopy within 2 years after primary surgery
  Interventions: Procedure: Patients with Cyclop lesion

INTERVENTIONS:
Procedure: Patients with Cyclop lesion — Arthroscopy with resection of Cyclop formation

SUMMARY:
Fibrous scar tissue formation (Cyclops) after a primary anterior cruciate ligament reconstruction (ACLr) may affect patients' ability to perform work and exercise to such an extent that further arthroscopic surgery may be necessary.

The purpose of the study is to estimate the 2-year incidence of removal of cyclops lesion after ACLr for a cohort of approximal 3000 patients operated at Aarhus University Hospital in the period 2005-2019.

Specifically, change in surgical technique and graft choice will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patient >18 years
* Primary ACL reconstruction

Exclusion Criteria:

* Multiligament reconstruction
* Revisions
* ACL reconstruction with double bundle graft

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary ACL reconstructed patients operated in the period 2005-2019
Sampling Method: Non-Probability Sample
Enrollment: 2556 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Cyclop lesion | 2 years
  Incidence of Arthroscopy with removal of Cyclop formation

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No